CLINICAL TRIAL: NCT03923829
Title: The Effect of Systemic Administration of Zinc on the Gingival Crevicular Fluid Level of Total Oxidant Capacity in Type 2 Diabetic Patients With Stage II and III Periodontitis After Non-surgical Periodontal Therapy
Brief Title: The Effect of Zinc on the Gingival Crevicular Fluid Level of Total Oxidant Capacity in Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulrahman Abdulqawi Awadh Abdulrab, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6653486
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Periodontitis
Keywords: zinc; Non-surgical Periodontal Therapy; stage II periodontitis; stage III periodontitis; gingival crevicular fluid; total oxidant capacity; Type 2 diabetic patients
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Zinc Sulfate; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and statistician will be blinded to the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc administration with scaling and root planing (Experimental): systemic administration of Zinc cap of 50 mg elemental zinc as zinc sulphate, once a day for 12 weeks in addition to scaling and root planing
  Interventions: Drug: Zinc Sulfate
- scaling and root planing (Active Comparator): scaling and root planing
  Interventions: Procedure: scaling and root planing

INTERVENTIONS:
Drug: Zinc Sulfate — systemic administration of Zinc sulfate with scaling and root planing
  Other Names: Zinc Sulfate with scaling and root planing
  Arms: Zinc administration with scaling and root planing
Procedure: scaling and root planing — scaling and root planing
  Arms: scaling and root planing

SUMMARY:
To evaluate the effect of systemic administration of zinc on the gingival crevicular fluid level of total oxidant capacity in controlled Type-2 diabetic patients with stage-II and III periodontitis after non-surgical periodontal therapy.

DETAILED DESCRIPTION:
Hypozincaemia and hyperzincuria is known to be present in patients with type-2 diabetes, and Zinc supplementation is known to be helpful in restoring plasma Zinc levels to normal,Zinc's deficiency can lead to an increase in circulating glucose due to beta cells malfunctioning and resistance to insulin, which makes it easier for type 2 diabetes mellitus (DM2) to happen ,Zinc was found to be a structural part of key anti-oxidant enzymes such as superoxide dismutase (SOD), and Zinc deficiency impaired their synthesis, leading to increased oxidative stress

ELIGIBILITY:
Inclusion Criteria:

* Controlled Type-2 diabetes mellitus
* Stage-II &III periodontitis
* At least 2 sites with clinical attachment loss 3 or 4 mm to ≥5 mm and radiographic bone loss 15% Extending to mid-third of root and beyond.
* Probing depth from ≤5 mm to ≥6 mm

Exclusion Criteria:

* Any periodontal or Antibiotic treatment during the last six months.
* Receiving trace element supplements in the previous three months
* Pregnant or lactating females
* Gastric or diuretic treatment
* Acute renal failure
* smoking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline Hb-A1c | change from baseline Hb-A1c at 3 monthes

SECONDARY OUTCOMES:
Hb-A1c | at the baseline and after 3 months
  Hb-A1c
Probing pocket depth | at the baseline and after 3 months
  Probing pocket depth Measured as the distance between the gingival margin and the apical part of the pocket will be measured using William's graduated periodontal probe.
Clinical attachment level | at the baseline and after 3 months
  It will be measured from the cemento-enamel junction till the apical part of the pocket.
Gingival index | at the baseline and after 3 months
  Gingival Index for a specific tooth == Average (points for the 4 surfaces)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Enji Ahmed, professor, Principal Investigator — Cairo University; Dr. weam elbattawy, Lecturer, Study Director — Cairo University; Dr. Ollfat Shaker, professor, Study Director — Cairo University

REFERENCES:
- [Result] Khan MI, Siddique KU, Ashfaq F, Ali W, Reddy HD, Mishra A. Effect of high-dose zinc supplementation with oral hypoglycemic agents on glycemic control and inflammation in type-2 diabetic nephropathy patients. J Nat Sci Biol Med. 2013 Jul;4(2):336-40. doi: 10.4103/0976-9668.117002. PMID 24082728
- [Result] Thomas B, Prasad RB, Shetty S, Vishakh R. Comparative Evaluation of the Lipid Profile in the Serum of Patients with Type II Diabetes Mellitus and Healthy Individuals with Periodontitis. Contemp Clin Dent. 2017 Jan-Mar;8(1):96-101. doi: 10.4103/ccd.ccd_1160_16. PMID 28566858